CLINICAL TRIAL: NCT02849717
Title: Pre-Habilitation Exercise Intervention for Patients Scheduled for Colorectal Surgical Resection
Brief Title: Pre-Habilitation Exercise Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Fergal Fleming, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 59142
Record Dates: First submitted 2016-07-19; First posted 2016-07-29 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Diseases; Colon Cancer; Rectal Cancer; Diverticular Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colonic Neoplasms; Rectal Neoplasms; Diverticular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (No Intervention): Subjects are advised to maintain their normal level of activity
- Home-Based Exercise (Active Comparator): Progressive walking and resistance exercise treatment
  Interventions: Behavioral: Exercise for Cancer Patients

INTERVENTIONS:
Behavioral: Exercise for Cancer Patients — a standardized, daily, home-based, progressive exercise program
  Other Names: EXCAP
  Arms: Home-Based Exercise

SUMMARY:
The purpose of this study is to see whether exercise can improve the health and well-being of patients scheduled to undergo surgery for a bowel related condition.

DETAILED DESCRIPTION:
The proposed randomized controlled trial aims to recruit 60 patients that have a primary diagnosis of either colon or rectal cancer, inflammatory bowl disease, or diverticular disease and are scheduled for elective surgery. This two-arm clinical trial of an intervention examining the efficacy of a home-based walking and progressive resistance exercise program for the relief of post-operative fatigue and improvement of functional outcome following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of one of the following: colon or rectal cancer, inflammatory bowel disease, or diverticular disease
* Be scheduled for elective (non- emergent) surgery
* Have the approval of their treating physician, study physician, or physician's designee to participate in maximal physiological fitness testing and a low to moderate home-based walking and progressive resistance exercise program.
* Be able to read English (since the assessment materials will be in a printed format).
* Be 18 years of age or older
* Give informed consent.

Exclusion Criteria:

* Have physical limitations (e.g. cardiorespiratory, orthopedic, central nervous system) that contraindicate participation in maximal physiological fitness testing, or a low to moderate home-based walking and progressive resistance program, as assessed by the Par-Q+ and clinician (or physician's designee)
* Must not be in active or maintenance stage of exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-03; Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for this study is fatigue assessed by the FACIT-F fatigue subscale.. | 12 weeks
  The primary analyses will involve examination of means, standard deviations, and effect sizes of the two arms on fatigue at all three times, separately by cohort and combined.

SECONDARY OUTCOMES:
Aerobic Capacity via VO2 maximum testing | 12 weeks
  The secondary aim is to provide preliminary data on the influence of a home-based walking and progressive resistance exercise program (EXCAP) plus standard care versus standard care alone on aerobic capacity in subjects who have undergone colorectal resection.
Skeletal Muscle Mass will be assessed using bio-electrical impedance assessment of muscle mass | 12 weeks
  The secondary aim is to provide preliminary data on the influence of a home-based aerobic and resistance exercise (EXCAP) intervention on skeletal muscle mass and its relationship to fatigue in subjects who have undergone colorectal resection.
Skeletal Muscle Mass will be assessed using CT assessment of muscle mass | 12 weeks
  The secondary aim is to provide preliminary data on the influence of a home-based aerobic and resistance exercise (EXCAP) intervention on skeletal muscle mass and its relationship to fatigue in subjects who have undergone colorectal resection.
Circulating Levels of Pro-Inflammatory Cytokines will be measured by standard Complete Blood Count (CBC) differential procedures. | 12 weeks
  The secondary aim is to provide preliminary data on the influence of a home-based aerobic and resistance exercise intervention (EXCAP) plus standard care versus standard care alone on the circulating levels of pro-inflammatory cytokines (IL-6, IL-8,IL-10, IL-1B,and IFN-y) and TNFr1 cytokine receptor expression in subjects who have undergone colorectal resection.
Post-operative Complications will be extracted from patient charts and will be classified for severity using the Clavien-Dindo classification of surgical complications. | 12 weeks
  The secondary aim is to provide preliminary data on the influence of a home-based walking and progressive resistance exercise program (EXCAP) plus standard care versus standard care alone on post-operative complications in subjects who have undergone colorectal resection.
Quality of Life (QOL) on self reported psychological distress questionnaires: Profile of Mood States (POMS). | 12 weeks
  The secondary aim is to provide preliminary data on the influence of a home-based walking and progressive resistance exercise program (EXCAP) plus standard care versus standard care alone on quality of life (QOL) in subjects who have undergone colorectal resection.
Quality of Life (QOL) on self reported psychological distress questionnaires: Spielberg State/Trait Anxiety Inventory (STAI Form Y-1). | 12 weeks
  The secondary aim is to provide preliminary data on the influence of a home-based walking and progressive resistance exercise program (EXCAP) plus standard care versus standard care alone on quality of life (QOL) in subjects who have undergone colorectal resection.

CONTACTS AND LOCATIONS:
Overall Officials: Fergal Fleming, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States